CLINICAL TRIAL: NCT01577394
Title: Oculomotor Recording in the Contribution to the Early Differential Diagnosis of Dementia With Lewy Bodies and Alzheimer's Disease
Brief Title: Oculomotor Testing in the Differential Diagnosis of Dementia
Acronym: OculoMacl
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM 09158
Record Dates: First submitted 2012-02-23; First posted 2012-04-13 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Lewy Body Disease; Alzheimer's Disease
Keywords: Alzheimer disease; Lewy Body Disease; Cognitive Disorders; Neurodegenerative Diseases; Differential diagnosis; Eye movement
MeSH Terms: conditions — Lewy Body Disease; Alzheimer Disease; Cognitive Dysfunction; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early stage of dementia (Experimental): oculomotor measurements
  Interventions: Other: oculomotor measurements

INTERVENTIONS:
Other: oculomotor measurements — The variability is indicated by the coefficient of variation (i.e. standard-error/mean) of saccades latencies in the gap paradigm.
  Mean reflexive saccades latency Percentage of express saccades
  Other Names: reflexive saccades latencies

SUMMARY:
The aim of this study is to determine whether saccadic eye movement recording may help in the discrimination between Lewy body dementia and Alzheimer disease, in the early stages of the disease.

Study type: Interventional Study design: Intervention Model: Single group assignment Primary purpose: Diagnostic

DETAILED DESCRIPTION:
Dementia with Lewy bodies (DLB) is the second most common cause of neurodegenerative dementia. In its early stages, the differential diagnosis of DLB and Alzheimer's disease (AD) can be challenging. The differential diagnosis is particularly important given that patients with DLB respond well to cholinesterase inhibitors but show sensitivity to neuroleptic medications which are contraindicated in DLB. DLB tends to progress more quickly than Alzheimer's disease. Diagnostic accuracy may be improved. Oculomotor recording, easy to perform could be helpful in order to identify and reliably assess fluctuating attention performance in DLB patients.

Main objective:

- to improve differential diagnosis between DLB and AD in the early stages of the disease with oculomotor measurements

Secondary objectives:

* to examine the association between the oculomotor records and neuropsychological examination assessing attention abilities and their fluctuations
* to evaluate the benefit of complementary neuropsychological tests in the distinction between DLB and AD cases
* to examine the relationship between hippocampal volume and neuropsychological examination in DLB cases
* to examine the diagnostic performance of MRI (Support Vector Machine) between DLB and AD
* to examine the interest of CSF alpha synuclein concentration to discriminate DLB from AD
* to assess at one year variations in oculomotor test scores and neuropsychological test scores Method and design Longitudinal multicenter study including 100 patients with a DLB or AD diagnosis. Clinical examination at one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over
* Patients with a diagnosis of probable DLB or AD according to the Consortium on DLB criteria (McKeith et al 2005) for Lewy bodies dementia and according to DSM IV and NINCDS- ADRDA criteria for AD or patients in whom there is diagnostic uncertainty between DLB and AD
* No major sensory deficits
* MMSE > 20
* Having signed an informed consent form

Exclusion Criteria:

* Parkinson syndrome progressing for more than one year regarding cognitive impairment
* Use of AchEIs medication
* Taking or having taken anti Parkinson drugs
* Neuroleptic drugs over the previous three months
* Contraindication for lumbar puncture (i.e. anticoagulant agents)
* Patients with Geriatric Depression Scale (GDS) > 10
* Taking medication that could impact dopamine transporter's measurement
* Contraindication for MRI examination
* Diseases involving the short-term survival (shorter than one year)
* Not fluent in French
* Major sensory deficits that could interfere with cognitive assessment (visual and auditory)
* Being under guardianship
* Absence of caregiver/informant to sign informed consent form
* Non health insurance affiliation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Variability of reflexive saccades latencies | at one year
  The variability is indicated by the coefficient of variation (i.e. standard-error/mean) of saccades latencies in the gap paradigm. The variability and mean latency are expected to be increased while the percentage of express latencies decreased in DLB patients

SECONDARY OUTCOMES:
Correlations between oculomotor records and neuropsychological examination assessing attention abilities and their fluctuations | at one year
  This indicator concerns the standard Bravais-Pearson correlations between saccades latencies values and scores in neuropsychological tests.
Potential correlations between hippocampal volume and neuropsychological examination in DLB cases | at one year
  This indicator concerns the standard Bravais-Pearson correlations between neuro-psychological test scores and the measures of hippocampal volume
Cerebral atrophy differences between DLB and AD using SVM (Support Vector Machine) method | at one year
  score differences between the two groups
Percentage of alpha synuclein in CSF to discriminate DLB from AD | at one year
  score differences between the two groups
Variations at one year in oculomotor test scores and neuropsychological test scores | at one year
  comparing baseline and follow-up performance separately for each group
Mean reflexive saccades latency | at one year
  test differences in mean reflexive saccades latency between the two groups
Percentage of express saccades | at one year
  test differences in proportion of express saccades between the two groups
Correlations between neuropsychological tests scores assessing attention abilities and variability of reflexive saccades latencies | at one year
  This indicator concerns the standard Bravais-Pearson correlations between attention abilities test scores and the coefficient of variation of reflexive saccades latencies

CONTACTS AND LOCATIONS:
Overall Officials: Marc Verny, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - Pitié-Salpetriere hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No